CLINICAL TRIAL: NCT06536582
Title: Nutrition as a Risk Factor and Predictor of Treatment Outcome With Plasma Rich Growth Factors for Shoulder Tendinopathy
Brief Title: Nutrition Impact on PRGF Treatment for Tendinopathy
Acronym: NUTRITENDON
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: NUTRITENDON; 5xmille 2021CUPC43C2200237000 (Other Grant/Funding Number: Italian Ministry of health); L1054 Ricerca corrente (Other Grant/Funding Number: Italian Ministry of health)
Record Dates: First submitted 2024-03-19; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Tendinopathy; Metabolic Alterations
Keywords: nutritional status; responder and non-responder patients; orthobiologics; Platelet rich growth factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal weight patients: 23 subjects with body mass index (BMI) between 18.5 and 25 therefore considered normal weight, who undergo treatment with PRGF.
  Interventions: Biological: Platelet rich growth factor injection (autologous product)
- Over weight patients: 23 subjects with BMI values that exceed the considered range normal weight, therefore with BMI>25, who undergo the PRGF treatment
  Interventions: Biological: Platelet rich growth factor injection (autologous product)

INTERVENTIONS:
Biological: Platelet rich growth factor injection (autologous product) — All patients will undergo two PRGF injections, one at recruitment and one 14 days after the first injection. The injection site will be the shoulder with tendinopathy.

SUMMARY:
Given the close correlation reported in the literature between onset and progression of tendon pathology in subjects affected by the alteration of metabolic disorders such as obesity, diabetes mellitus and lipidic metabolic alterations, with the present study the association between the nutritional state, metabolic profile and clinical outcome of patients following treatment with blood-derived orthobiological for shoulder tendinopathies will be evaluated.

The primary aim of this study is to identify the proportion of tendinopatic patients responsive and non-responsive to treatment with "Platelet rich growth factors" PRGF at six months follow up and the correlation with their nutritional status.

DETAILED DESCRIPTION:
This is a single-center, observational study with an additional procedure (extra blood sampling routine, food questionnaires, anthropometric measurements for the evaluation of nutritional status), prospective, uncontrolled.

Male and female patients, between 18 and 70 years old suffering from tendinopathy of the shoulder who undergo conservative regenerative medicine procedures with autologous PRGF material at the IRCCS Galeazzi-Sant'Ambrogio Hospital of Milan and participants in the observational study "Use of Patient- Reported Outcome Measures (PROMs), objective clinical assessments and biomolecular technologies for monitoring patients undergoing treatments regenerative medicine" [REGAIN] will be enrolled for this study.

46 patients will be needed:

1. 23 subjects with body mass index (BMI) between 18.5 and 25 therefore considered normal weight, who undergo treatment with PRGF;
2. 23 subjects with BMI values that exceed the considered range normal weight, therefore with BMI>25, who undergo the PRGF treatment.

The general aim of the present study is to evaluate the correlation between the nutritional status of patients, the characteristics of the orthobiological product used for the treatment of shoulder tendon pathology and clinical outcomes after one-step conservative regenerative medicine treatment with PRGF in order to identify the ideal nutritional conditions to obtain the best clinical outcome from this type of treatment.

The primary objective of this study is to identify the proportion of tendinopatic patients responsive and non-responsive to treatment with orthobiological "Platelet rich growth factors" PRGF at six month follow up and the correlation with their nutritional status. To this end, responsive patients and non-responsive will be identified on the basis of the results of the VAS, ASES, Quick Dash, SPADI, WOOS scores, and Work index.

The secondary objectives of the study will be:

1) to Identify the proportion of responsive and non-responsive patients presenting shoulder tendinopathy to treatment with orthobiological "Platelet rich growth factors" PRGF at two and twelve months follow up and the correlation with their nutritional status. For this purpose, responsive and non-responsive patients will be identified on the basis of the results of the VAS, ASES, Quick Dash, SPADI scores, WOOS, and Work index.

Characterization of the PRGF product used for the treatment of each patient that will occur by qualitative and quantitative analysis of the content in extracellular vesicles, analysis of a panel of cytokines, chemokines and growth factors linked to inflammation and correlated to the state nutritional information of patients (e.g. resistin, P-selectin, interleukins etc.).

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age ≥18 years and ≤ 70 years
* Patients presenting shoulder tendinopathy
* Signing of the Informed Consent of the Regain observational study
* Signature of informed consent of the present study.

Exclusion Criteria:

* Pregnancy (ascertained by self-declaration), breastfeeding
* Inability to follow the study protocol
* Heart, kidney, oncological disease
* Neuropsychiatric disease
* Other conditions that, at the discretion of the investigator or physician, exclude enrollement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients, between 18 and 70 years old suffering from shoulder tendinopathy undergoing a conservative regenerative medicine procedure with autologous PRGF at the IRCCS Galeazzi-Sant'Ambrogio Hospital of Milan and participants at the observational study "Use of patients- Reported Outcome Measures (PROM), objective clinical assessments and biomolecular technologies for monitoring patients undergoing treatments regenerative medicine" [REGAIN] will be enrolled for this study.
  46 patients will be needed:
  1. 23 subjects with body mass index (BMI) between 18.5 and 25 therefore considered normal weight, who undergo treatment with PRGF;
  2. 23 subjects with BMI values that exceed the considered range normal weight, therefore with BMI>25, who undergo the PRGF treatment.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Responder and non-responder patient identification at 6 months follow-up. | 0-24 months
  The primary objective of this study is to identify the proportion of responder and non-responder patients with shoulder tendinopathy to treatment with orthobiological "Platelet rich growth factors" PRGF at six month follow up. Responsive and non-responsive patients will be identified on the basis of the results of the VAS, ASES, Quick Dash, SPADI, WOOS scores, and Work index.
Identification of nutritional status of responder and non-responder patients: complete blood count | 0-24 months
  Complete blood count (cell number/dl)
Identification of nutritional status of responder and non-responder patients: blood glucose | 0-24 months
  Blood glucose (mg/dl)
Identification of nutritional status of responder and non-responder patients: Hemoglobin A1C (HbA1c) | 0-24 months
  Hemoglobin A1C (HbA1c): mmol/mol
Identification of nutritional status of responder and non-responder patients: urea | 0-24 months
  Urea: mg/dl
Identification of nutritional status of responder and non-responder patients: creatinine | 0-24 months
  Creatinine: mg/dl
Identification of nutritional status of responder and non-responder patients: siderosis | 0-24 months
  siderosis: ug/dl
Identification of nutritional status of responder and non-responder patients: tryglicerides | 0-24 months
  tryglicerides (mg/dl)
Identification of nutritional status of responder and non-responder patients: cholesterol | 0-24 months
  Cholesterol (mg/dl)
Identification of nutritional status of responder and non-responder patients: Cholesterol HDL | 0-24 months
  Cholesterol HDL (mg/dl)
Identification of nutritional status of responder and non-responder patients: Glutamate-oxaloacetate transaminase | 0-24 months
  Glutamate-oxaloacetate transaminase: (U/l)
Identification of nutritional status of responder and non-responder patients: Glutamate-pyruvate transaminase | 0-24 months
  Glutamate-pyruvate transaminase: (U/l)
Identification of nutritional status of responder and non-responder patients: gamma GT | 0-24 months
  Gamma GT: U/l
Identification of nutritional status of responder and non-responder patients: calcium | 0-24 months
  Calcium: mg/dl
Identification of nutritional status of responder and non-responder patients: Vitamin D (25 OH) | 0-24 months
  Vitamin D (25 OH): ng/ml
Identification of nutritional status of responder and non-responder patients: ferritin | 0-24 months
  Ferritin (ng/ml)
Identification of nutritional status of responder and non-responder patients: | 0-24 months
  C reactive protein: (mg/dl)
Identification of nutritional status of responder and non-responder patients: thyroid stimulating hormone (TSH) | 0-24 months
  thyroid stimulating hormone (TSH): uIU/ml
Identification of nutritional status of responder and non-responder patients: Insulin | 0-24 months
  Insulin: uU/ml
Identification of nutritional status of responder and non-responder patients: Folates | 0-24 months
  Folates (ng/ml)
Identification of nutritional status of responder and non-responder patients: vitamin B 12 | 0-24 months
  Vitamin B 12 (pg/ml)
Anthropometric measurement: weight | 0-24 months
  weight (kg) measurement
Anthropometric measurement: height | 0-24 months
  height (m) measurement
Anthropometric measurement: waist circumference | 0-24 months
  waist circumference (cm) measurement
Anthropometric measurement: arm circumference measurements | 0-24 months
  arm circumference measurements (cm)
Anthropometric measurement: biceps folds measurement | 0-24 months
  biceps folds measurement (mm)
Anthropometric measurement: triceps folds measurement | 0-24 months
  triceps folds measurement (mm)
Anthropometric measurement: subscapular folds measurement | 0-24 months
  subscapular folds measurement (mm)
Anthropometric measurement: suprailiac folds measurement | 0-24 months
  suprailiac folds measurement (mm)

SECONDARY OUTCOMES:
Responder and non-responder patient identification at 2 months follow-up. | 2-26 months
  The secondary objectives of the study will be:
  to Identify the proportion of patients with shoulder tendinopathy responsive and non-responsive to treatment with orthobiological "Platelet rich growth factors" PRGF at two months follow up. For this purpose, responsive and non-responsive patients will be identified on the basis of the results of the VAS, ASES, Quick Dash, SPADI scores, WOOS, and Work index.
Responder and non-responder patient identification at 12 months follow-up. | 12-36 months
  The secondary objectives of the study will be:
  to Identify the proportion of patients with shoulder tendinopathy responsive and non-responsive to treatment with orthobiological "Platelet rich growth factors" PRGF at twelve months follow up. For this purpose, responsive and non-responsive patients will be identified on the basis of the results of the VAS, ASES, Quick Dash, SPADI scores, WOOS, and Work index.
The Platelet rich growth factors "PRGF" product used for the treatment of each patient will be characterizated: extracellular vesicles count | 24-26 months
  extracellular vesicles count: number/ml
The PRGF product used for the treatment of each patient will be characterizated: extracellular vesicles marker quantification | 24-26 months
  Identification of extracellular vesicles markers: Arbitrary Fluorescence Unit
The PRGF product used for the treatment of each patient will be characterizated- quantitative analysis of cytokines: CXCL8 | 24-26 months
  Quantitative analysis of cytokines (CXCL8): pg/ml
The PRGF product used for the treatment of each patient will be characterizated- quantitative analysis of growth factors: G-CSF | 24-26 months
  Quantitative analysis of growth factors: G-CSF (pg/ml)
The PRGF product used for the treatment of each patient will be characterizated- quantitative analysis of resistin | 24-26 months
  Quantitative analysis of resistin: pg/ml
The PRGF product used for the treatment of each patient will be characterizated- quantitative analysis of P-selectin | 24-26 months
  Quantitative analysis of P-selectin: pg/ml

OTHER OUTCOMES:
VAS | 2-36 months
  VAS: Visual analogue scales for grading of pain. The VAS ranges from 0 (no pain) to 10 (worst pain) ((consists of a 10 cm line with 10 mm (0.01 cm) to each point of the scale and two end-points representing no pain and worst possible pain, where 0 = no pain, 1-3 = mild, 4-6 = moderate and 7-10 = severe pain))
ASES SCORE | 2-36 months
  ASES (American Shoulder and Elbow Surgeons) Score: ASES score ranges from 0 to 100, with 0 the lowest level of function and 100 the highest level of function
Quick Dash Score | 2-36 months
  Quick Dash (Disabilities of Arm, Shoulder and Hand) score. The possible score ranges from 0 to 100 points. 0 points represent a complete, unrestricted function of the upper extremities, while 100 points represent the greatest possible functional impairment.
SPADI scores | 2-36 months
  SPADI (Shoulder Pain and Disability Index) scores. It evaluates pain and functional activities. Pain scale: 0 = no pain and 10 = the worst pain imaginable. Disability scale: 0 = no difficulty and 10 = so difficult it requires help. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
WOOS Index | 2-36 months
  WOOS (Western Ontario Osteoarthritis of the Shoulder) index. 0% is the worst possible result and 100% is the best possible results.
WORC Index | 2-36 months
  The WORC (Western Ontario Rotator Cuff) Index, is a disease-specific quality of life questionnaire, evaluating the change in symptoms and functional ability, specific to a RC tendinopathy.
  Total final WORC scores can, therefore, range from 0% (lowest functional status level) to 100% (the highest functional status)

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided